## A Study of Peripheral Neuropathy Clinical Trial Experiences: Insights from Patients

Outlined below is the informed consent form intended for peripheral neuropathy patients who are prospective participants in <a href="Power Clinical Trial's">Power Clinical Trial's</a> observational clinical study.

Date: March 22, 2024

## Study Overview

We warmly invite you to join our research endeavor. Enclosed is a consent form detailing the study's purpose and the implications of your involvement. If you encounter any unfamiliar terms or phrases, please don't hesitate to reach out to our research team for clarification. We encourage you to take your time in deciding whether to participate and to ask any questions that may arise. Feel free to discuss the study with your loved ones, personal physician, trusted healthcare providers, or community members. Participation in this study is entirely voluntary, and there is no obligation to take part.

Exploring Peripheral Neuropathy: An Observational Study Overview

This study is designed to observe and comprehend various factors influencing your peripheral neuropathy clinical trial enrollment process and their impact on your ability to participate and complete the trial.

The collected data will be anonymized and analyzed to identify trends related to the experiences of peripheral neuropathy patients, which often contribute to suboptimal enrollment rates or low completion.

As this clinical study is observational, there will be no changes to your treatment upon participation.

This document serves as written confirmation of the discussions you've had with our site staff or recruitment coordinators. It can also be used as a reference during your participation in this clinical study.

Understanding the Purpose of Peripheral Neuropathy Research

Clinical trials often show a bias toward specific demographic groups, yet limited research exists to elucidate which trial attributes influence participation.

This study will gather diverse data on the clinical trial experiences of peripheral neuropathy patients to ascertain which factors hinder a patient's ability to enroll in or complete a trial.

Furthermore, it aims to analyze data from various demographic perspectives to identify recurring trends that could provide insights for future peripheral neuropathy patients.

What Are the Benefits of Participating in This Clinical Study?

By joining this observational clinical trial, you play a crucial role in advancing our understanding of how to better assist future peripheral neuropathy patients. The findings could lead to enhancements in participation rates and broaden the scope of future studies.

Understanding the Risks of Participating in This Observational Clinical Study

Engaging in clinical trials may necessitate alterations to your treatment routines, which inherently carry certain risks.

However, as this is an observational clinical study, there will be no modifications to your treatment regimen, thus eliminating any associated risks related to treatment changes.

Throughout the trial, online reporting and video calls with participating peripheral neuropathy patients are utilized. One potential risk in this process is the potential for data breaches.

With Power's clinical trials, this risk is mitigated. We ensure that data shared during these calls is securely encrypted. Call logs and electronic copies of consent forms are stored anonymously in a highly secure environment.

Distinguishing Features of This Study Compared to Other Peripheral Neuropathy Clinical Trials

Unlike many other trials, this study is not an interventional clinical trial.

In interventional clinical trials, peripheral neuropathy patients are typically required to undergo a specific treatment regimen, which may differ from their current treatment.

However, as this is an observational clinical trial, there will be no recommendations or changes to your treatment.

If you wish to explore other studies, you can search for <u>peripheral neuropathy studies</u> on clinicaltrials.gov or <u>peripheral neuropathy clinical trials</u> on Power's website.

You can expand your knowledge of clinical trials and their participation rates by exploring the following resources:

MacLennan, Demi L., Jennifer L. Plahovinsak, Rob J. MacLennan, and Carolynn T. Jones. "Clinical trial site perspectives and practices on study participant diversity and inclusion." *Clinical Pharmacology & Therapeutics* 113, no. 3 (2023): 670-679.

Meyer, Shelby, Henok G. Woldu, and Lincoln R. Sheets. "Sociodemographic diversity in cancer clinical trials: new findings on the effect of race and ethnicity." *Contemporary Clinical Trials Communications* 21 (2021): 100718.

## Responsibilities of Peripheral Neuropathy Patients in This Study

As a participant in this study, you will need to complete bi-weekly surveys lasting approximately 30 minutes each. Additionally, there will be quarterly check-in calls scheduled throughout the duration of the clinical trial.

To be eligible for participation, you must currently be enrolled in an interventional clinical trial. Your treatment plan and methodology prescribed by your primary care physician will remain unaffected if you decide to join this observational study.

Throughout the trial, if you have any concerns or questions, it is important to reach out to our staff for clarification and assistance.

Before enrolling in this clinical study, it is necessary to consult with your care team.

## **Participant Confirmation**

I have thoroughly reviewed the information provided above, and it has been verbally discussed with me. All inquiries I raised were addressed satisfactorily.

I acknowledge that my participation in this observational study is entirely voluntary, and I retain the right to withdraw at any point. Signing this document does not waive any of my legal rights.

I am aware that I will receive a copy of this consent form for my records. By affixing my signature below, I am indicating my willingness to take part in the clinical study.

| Printed Name of Participant | |
|---|---|
| Participant Signature | |
| Date | |
| Confirmation of Informed Consent D | Discussion |
| I confirm that I have extensively reviewed | the content of this form with the participant. |
| I ensure that the participant comprehends associated with this clinical trial for periph | • |
| Printed name of Person Conducting Information | med Consent Discussion |
| Person Conducting Informed Consent Dis | cussion Signature |
| Date | |